CLINICAL TRIAL: NCT06612944
Title: Prophylactic Intervention for Relapse Prevention Post-Allogeneic Transplantation in Very High-Risk MDS Patients Based on IPSS-M Stratification: A Single-Arm, Prospective, Single-Center Clinical Study
Brief Title: Prophylactic Intervention for Relapse Prevention Post-Allogeneic Transplantation in Very High-Risk MDS Patients Based on IPSS-M Stratification
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Clinical Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHSYXY-202405-IPSSM-MDS
Record Dates: First submitted 2024-09-23; First posted 2024-09-25 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Myelodysplastic Syndromes, Adult
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Group (Experimental)
  Interventions: Drug: Prophylactic Intervention for Relapse Prevention Post-Allogeneic Transplantation

INTERVENTIONS:
Drug: Prophylactic Intervention for Relapse Prevention Post-Allogeneic Transplantation — 1.1 AZA + BCL2 Inhibitor (Preferred Regimen) Subcutaneous injection of azacitidine at 32 mg/m² per day for 5 consecutive days, with a 28-day cycle; BCL2 inhibitor (VEN): 400 mg per day orally for one week (if combined with a CYP450 inhibitor, reduce to 100 mg per day).
  1.2 AZA (DEC) + DLI For patients with TP53 mutations or those who do not respond to VEN, subcutaneous injection of azacitidine at 32 mg/m² per day for 5 consecutive days, with a 28-day cycle; decitabine at 5 mg/m² per day for 5 consecutive days, with a 28-day cycle (preferred for those with TP53 mutations). For patients without the option for DLI, regimen 1.1 is recommended.
  DLI: Begins 3 months post-transplantation, starting with a dose of 1×10^5 CD3+ T lymphocytes for haploidentical transplants, with doses increasing every 4-6 weeks to 5×10^5 CD3+ T lymphocytes, 1×10^6 CD3+, and 5×10^6 CD3+ T lymphocytes; for full-matched transplants, the starting dose is 5×10^5 CD3+ T lymphocytes with dose escalations as above to 1×1

SUMMARY:
By collecting interventional clinical data to assess the survival and relapse conditions of patients post-transplantation and comparing them with historical data, the primary study endpoint is the 1-year and 2-year relapse-free survival (RFS) post-transplantation. This includes the time from the start of treatment until the documentation of disease progression (bone marrow smear blast cells > 5% or extramedullary relapse) or death due to any cause, whichever occurs first. This experiment aims to improve the post-transplant survival rates of MDS patients classified as very high risk under the IPSS-M stratification and to explore pathways to prevent relapse.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years, inclusive, both male and female. Diagnosed with MDS according to WHO criteria and classified as very high-risk by IPSS-M scoring. The patient must have a suitable hematopoietic stem cell donor for allogeneic transplantation: Related donors must be at least 5/10 matched for HLA-A, -B, -C, -DQB1, and -DRB1
2. Unrelated donors must be at least 8/10 matched for HLA-A, -B, -C, -DQB1, and -DRB1. Hematopoietic Cell Transplantation-Comorbidity Index (HCT-CI) score of ≤ 2. ECOG performance status of 0-2. Adequate liver, kidney, cardiac, and pulmonary functions as follows: Serum creatinine ≤ 1.5× upper limit of normal (ULN)
3. Cardiac function: Ejection fraction ≥ 50%
4. Baseline oxygen saturation > 92%
5. Total bilirubin ≤ 1.5× ULN
6. ALT and AST ≤ 2.0× ULN
7. Pulmonary function: DLCO (corrected for hemoglobin) ≥ 40% and FEV1 ≥ 50%. Patients must be capable of understanding and willing to participate in the study, and must sign an informed consent form.

Exclusion Criteria:

1. Failure to proceed with stem cell reinfusion after unsuccessful pre-transplant conditioning. History of previous hematopoietic stem cell transplantation (HSCT). ECOG performance status > 2. Hematopoietic Cell Transplantation-Comorbidity Index (HCT-CI) score ≥ 3. Any unstable systemic disease including, but not limited to: unstable angina, cerebrovascular accident or transient ischemic attack within the past 3 months, myocardial infarction within the past 3 months, congestive heart failure (New York Heart Association [NYHA] class ≥ III), post-pacemaker implantation requiring medication for severe arrhythmias, severe liver, kidney, or metabolic diseases
2. patients with pulmonary arterial hypertension. Active, uncontrolled infection: hemodynamic instability related to infection, new symptoms or signs of worsening infection, radiological evidence of new infectious foci, persistent fever without signs or symptoms that cannot exclude infection. Need for treatment for Grade ≥2 epilepsy, paralysis, aphasia, new cerebral infarction, severe brain trauma, dementia, Parkinson's disease, schizophrenia. HIV infection. Active hepatitis B (HBV) or hepatitis C (HCV) requiring antiviral treatment
3. patients at risk of HBV reactivation, indicated by positive hepatitis B surface antigen or core antibody without antiviral therapy for hepatitis B. Pregnant or breastfeeding women. Men and women of childbearing potential unwilling to use contraception during the treatment and for 12 months post-treatment. Allergic to intervention drugs such as azacitidine, decitabine, or venetoclax.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-12 (Actual); Primary Completion 2027-11-12 (Estimated); Study Completion 2028-11-12 (Estimated)

PRIMARY OUTCOMES:
RFS：relapse-free survival | 1 year
RFS：relapse- free survival | 2 year

SECONDARY OUTCOMES:
OS：overall survival | 1 year
OS：overall survival | 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided